CLINICAL TRIAL: NCT02165007
Title: HAPLOIDENTICAL HEMATOPOIETIC STEM CELL TRANSPLANTATION FOR CHILDREN WITH SICKLE CELL DISEASE AND THALASSEMIA USING CD34+ POSITIVE SELECTED GRAFTS
Brief Title: Haploidentical Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director- Center for Cancer and Immunology Research, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAPSICKLE
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell-thalassemia Disease; Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peripheral blood stem cell graft that are CD34+ selected (Experimental): peripheral blood stem cell graft that are CD34+ selected. All patients will undergo reduced intensity conditioning regimen which followed by infusion of a peripheral blood stem cell graft collected from haploidentical family donors that are CD34+ positively selected using the CliniMACS device and Sirolimus will be used for GVHD prophylaxis and given for 9 months post-transplant and then tapered off by one year (see intervention).
  Interventions: Drug: peripheral blood stem cell graft that are CD34+ selected

INTERVENTIONS:
Drug: peripheral blood stem cell graft that are CD34+ selected — The preparatory regimen will consist of Hydroxyurea from Days -50 to -22, Alemtuzumab from days -21 to -19 (test dose Alemtuzumab on day -22), Fludarabine days -8 to -4, Thiotepa Day -4, Melphalan day -3 to -2 (Table 4a). In patients with intolerance to or have received alemtuzumab in the prior 6 months, alemtuzumab will be replaced with rabbit ATG on days -10 through -7, followed by infusion of a peripheral blood stem cell graft collected from haploidentical family donors that are CD34+ positively selected using the CliniMACS device. Sirolimus will be used for GVHD prophylaxis and given for 9 months post-transplant and then tapered off by one year.
  Other Names: Reduced intensity conditioning; Sirolimus

SUMMARY:
The study is designed as a Pilot/Phase 1 trial of reduced intensity Haploidentical HSCT in patients with sickle cell disease and thalassemia. The purpose of the study is to assess the safety and toxicity of reduced intensity conditioning haploidentical hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Research subjects will undergo reduced intensity conditioning (Hydroxyurea, ATG, Fludarabine, Thiotepa, Melphalan) followed by infusion of a peripheral blood stem cell graft collected from haploidentical family donors that are CD34+ positively selected using the CliniMACS device. Sirolimus will be used for GVHD prophylaxis and given for 9 months post-transplant and then tapered off by one year

The use of the CliniMACS device for CD34 selection will be performed at CNMC through cross-reference of the master file for CliniMACS CD34+ Reagent by Milteyni Biotech (BB-MF 8061).

CliniMACs is an electromechanical device intended to isolate certain cell subsets from mixed cell populations. When used in combination with the CliniMACs CD34 reagent, it is possible to prepare extremely pure populations of CD34+ cells with upwards of 5 logs depletion of contaminating T cells within a closed and sterile system.

We intend to use this system to select cells from HLA haploidentical related donors who have been mobilized with G-CSF prior to stem cell collection. Since previous investigations of this strategy in adult patients have not translated into enhanced long term survival, we intend to limit this protocol to patients under the age of 22 as they have more rapid immune reconstitution.

ELIGIBILITY:
Inclusion Criteria:

* First allogeneic transplant
* Age up to 22 years
* Patients with severe sickle cell disease (stroke, elevated TCD velocities, >2 acute chest syndrome, ongoing chronic red cell transfusion > 6 months)
* Patients with transfusion dependent thalassemia and evidence of iron overload
* Patients must have a related donor that is HLA-matched at >/=4 of 8 but <8/8 HLA-A, -B, -C and -DRB1
* Cardiac function: Shortening fraction >25%; ejection fraction >40%
* Estimated creatinine clearance greater than 50 mL/minute
* Pulmonary function: DLCO ≥40% (adjusted for hemoglobin) and FEV1≥50% in patients 7 years and older with normal cognitive function and able to perform the test adequately. If not able to complete the testing a CT chest will be required., oxygen saturation>91%
* Liver function: direct (conjugated) bilirubin < 2x the upper limit of normal and ALT/AST < 2.5x the upper normal limit.
* Signed informed consent.

Exclusion Criteria:

* Life expectancy less than 6 months
* Patients with uncontrolled bacterial, viral or fungal infections (undergoing appropriate treatment and with progression of clinical symptoms) within 1 month prior to conditioning. Patients with febrile illness or suspected minor infection should await clinical resolution prior to starting conditioning.
* Pregnant or breastfeeding patients
* Patients seropositive for the human immunodeficiency virus (HIV)
* Patient with active Hepatitis B or C determined by serology and/or NAAT
* Active hepatitis, bridging fibrosis or cirrhosis on liver biopsy (biopsy required for patients on chronic transfusion therapy for > 1 year and evidence of iron overload with ferritin >1000 ng/mL)
* Patients with suitable 8/8 HLA matched related and unrelated donors
* Patients who have an intolerance to or have received alemtuzumab in the prior 6 months will be excluded from enrollment unless alemtuzumab is replaced with rabbit ATG in the conditioning regimen

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2015-01; Primary Completion 2024-01 (Actual); Study Completion 2024-10 (Actual)

PRIMARY OUTCOMES:
Incidence of transplant related adverse outcomes | 60 days
  The primary endpoint of this trial is safety. Transplant related adverse outcomes and non-hematological toxicity will be measured through Day +60 on this objective to include:
  * Non-hematological severe (Grade IV and V) organ specific toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0)
  * Rates of non-engraftment
  * Severe acute (Grade III-IV)
  * Veno-occlusive disease of the liver
  * Idiopathic pneumonia syndrome
  * Seizures/Posterior reversible encephalopathy syndrome (PRES)

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival upto 2 years

OTHER OUTCOMES:
Graft failure | 2 years
  Graft failure upto 2 years
Grades II-IV and III-IV acute GVHD | 180 days
  Grades II-IV and III-IV acute GVHD at day +180
Chronic GVHD | 1 year
  Chronic GVHD by 1 yea
Transplant-related mortality | 100 days
  Transplant-related mortality at Day+ 100
Viral infection rates | 6 months
  Viral infection rates at 6 months: Reactivation of CMV, Adenovirus and EBV detected on peripheral blood monitoring or any visceral disease with documented molecular studies for these viruses within the first six months post transplantation will be recorded
Lymphocyte reconstitution | 1 year
  Lymphocyte reconstitution upto 1 year post transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296